CLINICAL TRIAL: NCT03274063
Title: Gout Self-Monitoring Aiming to Reach Target Serum Urate (Gout-SMART): Feasibility Study of Supported Self-management of Gout in Secondary Care Patients Requiring Escalation of Urate Lowering Therapy
Brief Title: Gout Self-Monitoring Aiming to Reach Target
Acronym: Gout-SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Principal Investigator, Philip Riches, Consultant Rheumatologist & Honorary Senior Lecturer, University of Edinburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GoutSMART_NHSL_2YCR
Record Dates: First submitted 2017-08-30; First posted 2017-09-06 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Intervention Model Description: Participants will be randomised in a ratio of 2:1 to either supported self management or usual care.
Who Masked: Outcomes Assessor
Masking Description: Laboratory staff measuring biochemical traits will be blind to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supported self-management (Active Comparator): Escalation of urate lowering therapy will be supervised by clinical research team based on results of participant self-testing
  Interventions: Other: Supported self-management
- Usual care (Sham Comparator): Escalation of urate lowering therapy will remain the responsibility of the participants primary care physician.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Supported self-management — Participants will be supplied with urate self-testing kits. Participants will have a mobile phone application installed which will prompt the participant to perform urate self-testing, enable the clinical research team to advise on escalation of urate lowering therapy, and collect quality of life data .
  Arms: Supported self-management
Other: Usual care — Participants will have a mobile phone application installed which will allow the research team to collect quality of life data.
  Arms: Usual care

SUMMARY:
This study evaluates whether a supported self-management approach to gout is able to achieve target levels of serum urate, and better control of gout flares.

DETAILED DESCRIPTION:
Gout is the most common cause of inflammatory arthritis with recurrent gout flares a cause of reduced quality of life, work absence and disability. Effective treatments are widely available and yet many patients never achieve control of their disease. Resolution of gout attacks requires sustained lowering of the levels of serum urate, which in practise is seldom achieved. A supported self-management approach to gout has been developed which incorporates self-testing of urate levels and a smartphone application that will prompt participants to self-test and allow clinical researchers to titrate urate lowering therapies.

The feasibility of this approach will be evaluated in patients with gout referred to secondary care. Participants will be randomised 2:1 to the intervention or a control group. The intervention group will be offered supported self-management incorporating self-testing of serum urate. The control group will receive usual care from their primary care physician. The primary outcome will be the proportion of patients achieving levels of serum urate at or below 0.3mmol/l by 6 months. Participants will be followed up for a total of 12 months to assess the broader health and economic impact of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of gout (as per American College of Rheumatology criteria)
* Physician recommendation that escalation of urate lowering therapy with allopurinol or febuxostat is appropriate.
* Serum urate >0.36mm/L.
* Patient has a mobile phone and is able to install GoutSMART (Gout Self-monitoring Aiming to Reach Target urate) application.

Exclusion Criteria:

* Subject is unable to provide consent
* Severe renal failure (eGFR <30) or established liver disease
* Previous adverse reaction to allopurinol or febuxostat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip L Riches, FRCP PhD, Principal Investigator — University of Edinburgh/NHS Lothian
Locations (1):
- Western General Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available on request.
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by the principal investigator. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Derived] Riches PL, Alexander D, Hauser B, Kuske B, Krause A. Evaluation of supported self-management in gout (GoutSMART): a randomised controlled feasibility trial. Lancet Rheumatol. 2022 May;4(5):e320-e328. doi: 10.1016/S2665-9913(22)00062-5. Epub 2022 Mar 24. PMID 38294032

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supported Self-management | Usual Care
Started | 40 | 20
Completed | 36 | 18
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supported Self-management | Usual Care | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (15.0) | 52.6 (14.1) | 52.8 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 37 | 19 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 38 | 20 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 40 | 20 | 60
Tophi [Count of Participants; unit: Participants] — Percentage of participants with self-reported tophi
  Participants | 10 | 6 | 16
Urate [Mean (Standard Deviation); unit: mmol/L] | 0.47 (0.07) | 0.51 (0.10) | 0.48 (0.09)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Target Urate Levels (24 Weeks)
Description: Percentage of participants achieving serum urate level at, or below, 0.3mmol/l
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-management | Usual Care
Number analyzed (Participants) | 40 | 20
Participants | 29 | 3

2. Secondary Outcome: Proportion of Participants Achieving Target Urate Levels (52 Weeks)
Description: Proportion of participants achieving serum urate level at, or below, 0.3mmol/l
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-management | Usual Care
Number analyzed (Participants) | 40 | 20
Participants | 32 | 9

3. Secondary Outcome: Flare Frequency
Description: Number of self-reported gout flares (months 7 to 12)
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: number of self-reported gout flares
Arm/Group | Supported Self-management | Usual Care
Number analyzed (Participants) | 36 | 18
number of self-reported gout flares | 0.81 (1.06) | 2.06 (2.6)

4. Secondary Outcome: Presence of Tophi
Description: Percentage of participants with tophi at 52 weeks
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supported Self-management | Usual Care
Number analyzed (Participants) | 36 | 18
Participants | 8 | 5

5. Secondary Outcome: EQ-5D-5L Quality of Life Score
Description: EQ-5D-5L (EuroqQol-5 level-5 dimension) self-reported quality of life score. Maximum score of 100 represents best possible health, minimum score of 0 represents worst possible health.
Time Frame: 52 weeks
Population: Recording of quality of life data was incomplete in this study and only available at close in the number of participants shown. This limitation is acknowledged in the published article of this trial
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supported Self-management | Usual Care
Number analyzed (Participants) | 36 | 8
units on a scale | 83.4 (11.1) | 79.1 (12)

6. Secondary Outcome: Work Absences
Description: Number of days lost at work due to gout flare
Time Frame: 52 weeks
Population: Measure available only in participants completing study
Measure: Mean (Standard Deviation); unit: number of work days lost
Arm/Group | Supported Self-management | Usual Care
Number analyzed (Participants) | 36 | 18
number of work days lost | 0.24 (1.35) | 0.11 (0.47)

7. Secondary Outcome: Healthcare Utilisation
Description: Number of scheduled and unscheduled medical appointments
Time Frame: 52 weeks
Population: Measure available only in participants completing study
Measure: Mean (Standard Deviation); unit: Number of medical appointments
Arm/Group | Supported Self-management | Usual Care
Number analyzed (Participants) | 36 | 18
Number of medical appointments | 0.083 (0.37) | 0.67 (1.08)

8. Secondary Outcome: Self-reported Medication Compliance (24 Weeks)
Description: Number of doses of medication omitted in preceding 2 weeks by self-report at 24 weeks.
Time Frame: 24 weeks
Population: Measure available only in participants completing study
Measure: Mean (Standard Deviation); unit: Number of doses missed
Arm/Group | Supported Self-management | Usual Care
Number analyzed (Participants) | 36 | 18
Number of doses missed | 0.57 (1.63) | 1.32 (2.63)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Supported Self-management | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/40 | 4/20
Other Adverse Events (participants affected / at risk) | 7/40 | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supported Self-management (N=40) | Usual Care (N=20)
Cardiovascular accident (Vascular disorders) | 1 (1) | 0 (0)
Hip replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bowel cancer (Gastrointestinal disorders) | 1 (1) | 0 (0)
skull fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supported Self-management (N=40) | Usual Care (N=20)
abdo pain (Gastrointestinal disorders) | 5 (5) | 1 (1)
skin rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT03274063/Prot_SAP_000.pdf